CLINICAL TRIAL: NCT01309919
Title: Bleeding Patterns and Complications After Postpartum Intrauterine Device (IUD) Placement: a Pilot Study
Brief Title: Bleeding Patterns and Complications After Postpartum IUD Placement: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baystate Medical Center (Other)
Responsible Party: Principal Investigator, Katharine White, Chief, Division of General OB/GYN, Baystate Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BH10-190
Record Dates: First submitted 2011-03-04; First posted 2011-03-07 (Estimated); Results first posted 2015-01-29 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Postpartum Period
Keywords: intrauterine device; Mirena; levonorgestrel intrauterine system; postpartum contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IUD Arm (Active Comparator): Subjects who receive an IUD within 48 hours of delivery (vaginal or cesarean birth)
  Interventions: Device: IUD; Other: Diary
- Diary Arm (Other): Subjects who will not have an IUD placed postpartum; they may use another form of contraception, or no form at all
  Interventions: Other: Diary

INTERVENTIONS:
Device: IUD — Placement of the IUD after delivery (vaginal or cesarean birth), either immediately (within 10 minutes of placental delivery) or delayed (within 48 hours of delivery). Subjects will also keep a bleeding diary for three months postpartum.
  Other Names: Mirena intrauterine system
  Arms: IUD Arm
Other: Diary — Subjects will keep a bleeding diary for three months
  Other Names: bleeding diary (three-month calendar)

SUMMARY:
The purpose of the study is to determine the feasibility of placing the levonorgestrel-releasing intrauterine system (LNG - IUS, Mirena®) post-delivery. The investigators will gain information about complications at the time of placement; the investigators will also examine the expulsion rate, side effects, bleeding patterns and subject satisfaction at various time periods after insertion.

DETAILED DESCRIPTION:
This trial is a prospective two-arm cohort study to examine feasibility, complications, and patient satisfaction related to postpartum IUD placement, to be conducted at Baystate Medical Center (BMC).

There are two groups in this study. The first group is women who choose to have an IUD placed after delivery at BMC (IUD arm). The second group is women who decline an IUD but who will complete bleeding diaries for six-months postpartum (diary arm). We chose the LNG-IUS due to its high patient satisfaction rates and variety of non-contraceptive benefits.

The standard of care for postpartum contraception is to provide women with information about her choices during her pregnancy, and to provide her with a method at hospital discharge after delivery. We will approach women at their routine prenatal visits. Women will be counseled by their provider about the risks, benefits and alternatives of all of the available methods of birth control (pills, patch, ring, injection, implant, IUD and sterilization). We will provide written information about her choices. We will discuss in detail the issues surrounding postpartum IUD placement, which most women will not be familiar with as an option, and provide a detailed information sheet for her to take home. We will revisit the issue of contraception at each subsequent visit until the patient has made a decision about what method she wishes to use.

IUD ARM

All women who request postpartum IUD placement will be offered enrollment in the study in the IUD arm. If a patient wishes to enroll, we will obtain written informed consent for the study and the LNG-IUS. We will administer a brief demographic and contraceptive history questionnaire. Subjects will be given a prescription for the LNG-IUS to bring with them to the hospital at the time of their delivery. A notation about study involvement will be made in the problem list of the subject's electronic prenatal record, and she will be reminded by her provider at each subsequent visit to bring the IUD when she comes to the hospital for delivery.

The Mirena IUS (Bayer Pharmaceuticals) is a sterile, levonorgestrel-releasing (20 mcg/day) intrauterine system indicated for intrauterine contraception for up to 5 years. The local mechanism by which continuously released levonorgestrel enhances contraceptive effectiveness of Mirena has not been conclusively demonstrated. Studies of Mirena prototypes have suggested several mechanisms that prevent pregnancy: thickening of cervical mucus preventing passage of sperm into the uterus, inhibition of sperm capacitation or survival, and alteration of the endometrium.

All LNG-IUS insertions will be performed by the PI or by 2nd year obstetrics and gynecology residents. These residents all have experience with traditional IUD insertions, and they will be trained by the PI in postpartum IUD insertion. Training will involve a short lecture, practice insertions on a pelvic model, then observing a postpartum insertion by the PI. Insertions will be performed at one of three times:

1. at the time of vaginal delivery, within 10 minutes of placental delivery (immediate placement);
2. at the time of cesarean delivery, within 10 minutes of placental delivery (immediate placement);
3. within 48 hours of either vaginal delivery or cesarean delivery (delayed placement).

At the time of vaginal delivery, the LNG-IUS will be inserted guided by trans-abdominal ultrasound to help ensure placement as close to the fundus as possible. If ultrasound is unavailable, another attempt at IUD placement will be made when the ultrasound becomes available.

At the time of cesarean delivery, the LNG-IUS will be placed prior to closure of the uterine incision.

At the time of delayed placement, subjects will be offered a dose of their routine postpartum pain medication (ibuprofen or oxycodone) prior to insertion. The LNG-IUS will be inserted guided by trans-abdominal ultrasound to help ensure placement as close to the fundus as possible. If ultrasound is unavailable, another attempt at IUD placement will be made when the ultrasound becomes available.

If a subject has not filled the prescription for the IUD by the time of delivery, we will submit an electronic prescription to the hospital pharmacy for the IUD, and the IUD may be picked up by a family member or friend and brought to L&D for placement. If a subject has left the IUD at home when she comes into the hospital for delivery, the IUD may be brought into the hospital by a family member or friend; if the IUD arrives at the hospital after delivery, she will be scheduled for a delayed postpartum placement. If the subject has been unable to obtain the IUD by 48 hours after delivery, she will be offered interval placement at the time of her postpartum visit.

All subjects will receive a bleeding diary to complete at home. We will call subjects at two weeks postpartum. During this telephone call we will ask questions regarding short term complications such as bleeding and signs of infection. If the subject has seen a medical professional before this phone call, or the LNG-IUS was expelled or removed, specific questions will be asked regarding these circumstances. At their six week postpartum visit, subjects will review their bleeding diary with study staff, complete a questionnaire and be evaluated for intrauterine IUD placement. If the tail strings are not visible a trans-vaginal ultrasound will be performed to assess placement. An intra-cervical LNG-IUS will be considered an expulsion and removal will be performed. Subjects will be counseled to return to clinic if they suspect expulsion at any time. We will provide stamped envelopes for subjects to mail back their bleeding diary at 12 weeks postpartum. We will call subjects at 12 weeks and six months postpartum regarding complications and specific questions about their satisfaction with the LNG-IUS.

DIARY-ONLY ARM

Women who do not want a postpartum IUD but who are interested in study participation will be offered enrollment in the diary-only arm. If a patient wishes to enroll, we will obtain written informed consent for the study and we will administer a brief demographic and contraceptive history questionnaire. Subjects will be given the bleeding diary to start after their discharge from the hospital after delivery. We will provide stamped envelopes for subjects to mail back their bleeding diary at 12 weeks postpartum.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* speak either English or Spanish
* desire to use an IUD as their postpartum contraception (IUD arm)
* do NOT desire an IUD as their contraception (Diary Only arm)
* plan to deliver at Baystate Medical Center.

Exclusion Criteria:

* history of sexually transmitted infection during the three months prior to enrollment
* desiring of another pregnancy within six months of giving birth
* routine contraindications to IUD:
* cavity-distorting uterine fibroids or uterine anomalies
* known or suspected uterine or cervical neoplasia
* acute liver disease or liver tumor
* history of breast cancer

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katharine O White, MD, MPH, Principal Investigator — Baystate Medical Center
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intrauterine Device (IUD) Arm: Subjects who receive an IUD within 48 hours of delivery (vaginal or cesarean birth)
  IUD: Placement of the IUD after delivery (vaginal or cesarean birth), either immediately (within 10 minutes of placental delivery) or delayed (within 48 hours of delivery). Subjects will also keep a bleeding diary for three months postpartum.
  Diary: Subjects will keep a bleeding diary for three months
Period: Overall Study
Arm/Group | Intrauterine Device (IUD) Arm | Diary Arm
Started | 75 | 75
Completed | 58 | 27
Not Completed | 17 | 48
Not completed — Did not receive a postpartum IUD | 17 | 48

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IUD Arm | Diary Arm | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (5) | 24 (5) | 24.5 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 75 | 150
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47 | 38 | 85
  Not Hispanic or Latino | 27 | 37 | 64
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  White | 53 | 49 | 102
  Black | 8 | 14 | 22
  Other | 14 | 12 | 26
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 32.4 (7) | 31.6 (7) | 32 (7)

OUTCOME MEASURES:

1. Primary Outcome: Bleeding Patterns
Description: Number of bleeding and spotting days in the first six weeks and subsequent six weeks postpartum
Time Frame: 12 weeks post-partum
Population: We were able to analyze all returned bleeding diaries (25 participants in IUD Arm, 27 participants in Diary Arm)
Measure: Median (Full Range); unit: days
Arm/Group | IUD Arm | Diary Arm
Number analyzed (Participants) | 25 | 27
days
  First 6 wks PP - Bleeding | 15 [6 to 42] | 18 [8 to 42]
  First 6 wks PP - Spotting | 13 [0 to 29] | 7 [0 to 33]
  Second 6wks PP - Bleeding | 5.5 [0 to 42] | 8 [0 to 42]
  Second 6wks PP - Spotting | 7.5 [0 to 42] | 4 [0 to 30]

2. Secondary Outcome: Expulsions
Description: Incidence of spontaneous IUD expulsion in the six months after insertion
Time Frame: 6 months
Population: We assessed the number of expelled IUDs for all participants who had an IUD placed
Measure: Number; unit: participants
Arm/Group | IUD Arm | Diary Arm
Number analyzed (Participants) | 58 | 0
participants | 3 |

3. Secondary Outcome: Satisfaction
Description: Participant satisfaction with the IUD at 12 weeks post-insertion
Time Frame: 12 weeks post-partum
Population: We assessed satisfaction with the IUD of all participants who completed the 12-week follow up call
Measure: Number; unit: % of participants who received an IUD
Arm/Group | IUD Arm | Diary Arm
Number analyzed (Participants) | 44 | 0
% of participants who received an IUD
  Very satisfied | 82 |
  Somewhat satisfied | 11 |

4. Secondary Outcome: Insertion Time
Description: Time of insertion of the IUD
Time Frame: immediate
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | IUD Arm | Diary Arm
Number analyzed (Participants) | 58 | 0
minutes | 5.5 (4.3) |

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 6 months
Arm/Group | IUD Arm | Diary Arm
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 0/75 | 0/75

LIMITATIONS AND CAVEATS:
Low rate of bleeding diary return limited our assessment of the primary outcome of bleeding/spotting days after delivery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes